CLINICAL TRIAL: NCT01245478
Title: Clinical Outcome and 5-year Implant Survival Rate Among Adult Revision Total Knee Arthroplasty Patients With DePuy Implant Components
Brief Title: DePuy Revision TKA Implant 5yr Survivorship
Status: Withdrawn | Type: Observational
Why Stopped: Retrospective record review only (no subject enrollment). Contract never executed between Sponsor and Site.
Sponsor: The New England Baptist Hospital (Other)
Collaborators: Depuy, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IIS-000105
Record Dates: First submitted 2010-11-19; First posted 2010-11-22 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Complications; Arthroplasty, Mechanical
Keywords: Surgical Procedures, Elective

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This will be a retrospective chart review of 200 charts of adult patients who have undergone a revision TKA at New England Baptist Hospital and who received implant component(s) manufactured by DePuy Orthopedics. The data will be collected retrospectively after patients are seen clinically for a minimum of five years after surgery to answer:

1. What is the five-year survivorship of revision a knee prosthesis containing components manufactured by DePuy Orthopedics among adult revision TKA patients?
2. What patient factors are associated with the need for re-operation after revision TKA among patients receiving DePuy implant components? How do clinical outcomes change from baseline over the five-year follow-up after revision TKA surgery?

Data collection will include patient-reported and clinician-reported measures.

ELIGIBILITY:
Inclusion Criteria:

* Received a Revision TKA (must have been initial revision)

  --Received J&J/DePuy implant components for initial revision
* Procedure performed at New England Baptist Hospital

Exclusion Criteria:

* 2nd Revision TKA on knee
* Received femoral or tibial components not of DePuy manufacture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any NEBH patients who received DePuy implant components during a Revision TKA procedure, performed by either:
  * Dr. Geoffrey Van Flandern
  * Dr. David Mattingly
  * Dr. James Nairus
  * Dr. James Bono
  * Dr. Daniel Ward
  * Dr. Carl Talmo
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-11; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Richmond, MD, Principal Investigator — New England Baptist Hospital